CLINICAL TRIAL: NCT07212049
Title: Using Ultrasound as an Alternative to Radiography in Measuring Magnetically Controlled Growing Rods (MCGR) in Tibia and Femur Lengthening Patients
Brief Title: Ultrasound Use to Measure Magnetically Controlled Growing Rods
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Jason Malone, Pediatric Orthopedic Surgeon, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2169786
Record Dates: First submitted 2025-09-08; First posted 2025-10-21 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Limb Length Discrepancy
Keywords: limb lengthening; leg length difference
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasound of lengthening rod (Experimental): All patients will have an ultrasound measuring the lengthen of the internal rod
  Interventions: Device: ultrasound measurement; Diagnostic Test: X-ray imaging of tibia and/or femur

INTERVENTIONS:
Device: ultrasound measurement — Three different measurements will be obtained using an ultrasound to determine the length gained from lengthening the tibia and/or femur with an internal lengthening rod. Please see the protocol on the locations that will me measured.
Diagnostic Test: X-ray imaging of tibia and/or femur — All patients will have an x-ray with two views anterior-posterior and lateral to measuring the lengthening of the internal rod. Please see the protocol for locations of the measurements being obtained.
  Other Names: Radiographs

SUMMARY:
The goal of this clinical trial is to learn if an ultrasound can measure the length of an internal tibia and femur lengthening rod. The main questions it aims to answer are:

Can an ultrasound be used to measure the length of an internal magnetic lengthening nail in a tibia or femur? Can an ultrasound measure the rod lengthening as well as an ultrasound? Researchers will compare the length of an internal magnetic lengthening rod with both x-rays and ultrasound

Participants will:

Have standard x-rays every week They will also have an ultrasound of the femur or tibia

DETAILED DESCRIPTION:
Limb lengthening with expanding intramedullary rods has become the standard of care for limb lengthening procedures. The procedure entails performing an osteotomy of the short bone and placing a mechanical expanding intramedullary nail. The aim of the study is to explore the role of ultrasound to measure tibia and femur lengthening procedures and compare the accuracy to standard radiographs.

The study design is a prospective, pilot study of 5 tibias and 5 femurs. Measurements of the femurs and tibias will be obtained in 3 separate locations to try to identify areas that can be visualized and measured by an ultrasound. The cost of the ultrasound will be compared to the cost of x-rays, and any pain regarding imaging modalities will also be compared

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing tibia or femur lengthening with an intramedullary mechanical rod.

Exclusion Criteria:

* Patients who underwent lengthening procedure with any other device such as external fixator.
* Patients under 8 years old and over 21 years of age

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Measurement of the lengthening rod | Once a week during the lengthening process, up to 10 weeks
  ultrasound measurement of the length of the internal lengthening rod
X-ray measurement of the lengthening rod | Once a week during the lengthening process, up to 10 weeks
  X-ray measurement of the internal lengthening rod at three points on the rod.

SECONDARY OUTCOMES:
Cost of imaging | Once a week during the lengthening process, up to 10 weeks
  The cost of ultrasound and x-rays. The ultrasound has no cost as it is a point-of-care device. The x-ray cost will derived from the mast charge that is post online for Nemours Children's Hospital Florida. The cash charge for a tibia two view x-ray is $471. The cash charge for a femur two view x-ray is $282.
Pain reported during imaging | Once a week during the lengthening process, up to 10 weeks
  Pain experienced will measured with Wong-Baker faces pain rating scale during imaging with x-ray and ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Hospital Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stokes OM, O'Donovan EJ, Samartzis D, Bow CH, Luk KD, Cheung KM. Reducing radiation exposure in early-onset scoliosis surgery patients: novel use of ultrasonography to measure lengthening in magnetically-controlled growing rods. Spine J. 2014 Oct 1;14(10):2397-404. doi: 10.1016/j.spinee.2014.01.039. Epub 2014 Jan 31. PMID 24486476
- [Background] Cobanoglu M, Shah SA, Gabos P, Rogers K, Yorgova P, Neiss G, Grissom L, Mackenzie WG. Comparison of Intended Lengthening of Magnetically Controlled Growing Rods: Ultrasound Versus X-Ray. J Pediatr Orthop. 2019 Feb;39(2):e141-e146. doi: 10.1097/BPO.0000000000001072. PMID 29016427
- [Background] Yoon WW, Chang AC, Tyler P, Butt S, Raniga S, Noordeen H. The use of ultrasound in comparison to radiography in magnetically controlled growth rod lengthening measurement: a prospective study. Eur Spine J. 2015 Jul;24(7):1422-6. doi: 10.1007/s00586-014-3589-z. Epub 2014 Sep 26. PMID 25256680
- [Background] Cheung JP, Bow C, Samartzis D, Ganal-Antonio AK, Cheung KM. Clinical utility of ultrasound to prospectively monitor distraction of magnetically controlled growing rods. Spine J. 2016 Feb;16(2):204-9. doi: 10.1016/j.spinee.2015.10.044. Epub 2015 Oct 30. PMID 26523963
- [Background] Schiedel FM, Buller TC, Rodl R. Estimation of patient dose and associated radiogenic risks from limb lengthening. Clin Orthop Relat Res. 2009 Apr;467(4):1023-7. doi: 10.1007/s11999-008-0624-6. Epub 2008 Nov 22. PMID 19030942
- [Background] Laubscher M, Mitchell C, Timms A, Goodier D, Calder P. Outcomes following femoral lengthening: An initial comparison of the Precice intramedullary lengthening nail and the LRS external fixator monorail system. Bone Joint J. 2016 Oct;98-B(10):1382-1388. doi: 10.1302/0301-620X.98B10.36643. PMID 27694593

DOCUMENTS (6):
  • Study Protocol and Statistical Analysis Plan (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT07212049/Prot_SAP_000.pdf
  • Informed Consent Form: 7-11 year old Consent Guardian Assent (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT07212049/ICF_001.pdf
  • Informed Consent Form: 12 to 17 year old assent (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT07212049/ICF_002.pdf
  • Informed Consent Form: 7-11 year old Consent Guardian (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT07212049/ICF_003.pdf
  • Informed Consent Form: consent for adult (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT07212049/ICF_004.pdf
  • Informed Consent Form: 12 to 17 year old Guardian concent (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT07212049/ICF_005.pdf